CLINICAL TRIAL: NCT04355403
Title: A Prospective, Randomized, Controlled, Open-label Clinical Investigation to Assess the Performance and Safety of Hyalo Gyn Gel Prefilled Applicators on the Treatment of Vaginal Atrophy in Postmenopausal Women
Brief Title: Performance and Safety of Hyalo Gyn Gel on the Treatment of Vaginal Atrophy in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QQ53-18-01
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Vulvovaginal Atrophy
Keywords: Hyaluronic Acid; Post-menopause

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyalo Gyn gel (Experimental): Vaginal application of Hyalo Gyn gel in prefilled applicators
  Interventions: Device: Hyalo Gyn gel in prefilled applicators
- No treatment (No Intervention): No treatment application

INTERVENTIONS:
Device: Hyalo Gyn gel in prefilled applicators — One vaginal application of Hyalo Gyn gel every 3 days to a total of 12 consecutive weeks.
  Arms: Hyalo Gyn gel

SUMMARY:
This clinical investigation evaluates the performance and safety of Hyalo Gyn, a hyaluronic acid derivative based vaginal gel for the treatment of symptoms of vulvo-vaginal atrophy in post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman (≥12 months since last spontaneous menstrual period, or having 6 months of spontaneous amenorrhea with serum FSH levels >40 IU/L), both natural postmenopause or medical postmenopause (breast cancer patients undergoing a concurrent treatment with aromatase inhibitors or tamoxifen).
* Women between 18 and 75 years of age.
* Vaginal pH ≥5.
* Vulvovaginal atrophy with VHI < 15.
* At least one of the following symptoms of vulvar and vaginal atrophy, assessed as moderate to severe: vaginal dryness, vaginal and/or vulvar irritation/ itching, dysuria, vaginal pain associated with sexual activity.
* Women with active sex life.
* Patients who give written informed consent to participate in the trial.

Exclusion Criteria:

* Treatment with another investigational product within the previous 3 months.
* Previous participation in any clinical study with Hydeal-D based investigational products.
* Patients in previous treatment with any kind of no-hormonal products for local treatment of vaginal atrophy within 1 week
* Patients in previous treatment with either oral or topical hormonal products within 1 month.
* Patients that present clinical signs of vaginal infections such as trichomonas, candida, and bacterial vaginosis (BV); history of vulvovaginal contact allergy or with a diagnose of vulvovaginal lichen.
* Patients with acute hepatopathy, embolic disorders, severe primary disease of the kidney and hematopoietic system, and history of malignant tumors.
* Positive history of hypersensitivity hyaluronic acid or to any component of the medical device.
* Any condition in the investigator's opinion not suitable for the inclusion of the patient.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Selection of post-menopausal women with symptoms of vulvovaginal atrophy
Enrollment: 80 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Change of patient's perception of vulvovaginal dryness | From baseline to 12 weeks of treatment
  Change of patient's perception of vulvovaginal dryness associated with vulvovaginal atrophy in postmenopausal women in Hyalo Gyn gel group compared to no-treatment group. The vulvovaginal dryness was reported on a four-point scale (0=absent, 1=mild, 2=moderate, 3=severe).

SECONDARY OUTCOMES:
Change of patient's perception of vulvovaginal dryness | From baseline to 4 weeks of treatment
  Change of patient's perception of vulvovaginal dryness associated with vulvovaginal atrophy in postmenopausal women in Hyalo Gyn gel group compared to no-treatment group. The vulvovaginal dryness was reported on a four-point scale (0=absent, 1=mild, 2=moderate, 3=severe).
Change of patient's perception of vulvovaginal symptoms | From baseline to 4 and 12 weeks of treatment
  Change of patient's perception of symptoms associated with vulvovaginal atrophy in postmenopausal women in Hyalo Gyn gel group compared to no-treatment group. Each symptom (dryness, irritation/itching, soreness, dysuria, dyspareunia) will be reported on a four-point scale (0=absent, 1=mild, 2=moderate, 3=severe)
Change of the average score of Vaginal Health Index (VHI) | From baseline to 4 and 12 weeks of treatment
  Change of VHI in postmenopausal women in Hyalo Gyn gel group compared to no-treatment group. VHI will be calculated on the basis of vaginal elasticity, vaginal fluid volume, vaginal pH, vaginal mucosa epithelial integrity, and vaginal moisture on a scale ranging from 1 (poorest) to 5 (best). VHI assigned score is the sum of subscores and ranges from 5 to 25. A lower score corresponds to a greater atrophy.
Change of vaginal pH | From baseline to 4 and 12 weeks of treatment
  Change of vaginal pH in postmenopausal women in Hyalo Gyn gel group compared to no-treatment group. The pH values are grouped on a four-point scale and scored respectively: pH lower than 5 = 0; pH between 5 and 5.49 = 1; pH between 5.5 and 6.49 = 2; pH higher than 6.49 =3.
Improvement of sexual function through questionnaire Female Sexual Function Index (FSFI) | From baseline to 4 and 12 weeks of treatment
  Improvement of sexual function in postmenopausal women in Hyalo Gyn gel group compared to no-treatment group. Female Sexual Function Index (FSFI) questionnaire consists of six domains - desire (two items), arousal (four items), lubrication (four items), orgasm (three items), satisfaction (three items), and pain (three items) - answered on a five-point Likert scale (0, no sexual activity; 1, never/very low; 5, always/very high). A score is calculated for each of the six domains, and the total score is obtained by summing all of the items. Total score ranges from 2 to 36. A lower score corresponds to a greater sexual dysfunction.
Improvement of sexual function through questionnaire Female Sexual Distress Scale-Revised (FSDS-R) | From baseline to 4 and 12 weeks of treatment
  Improvement of sexual function in postmenopausal women in Hyalo Gyn gel group compared to no-treatment group. Female Sexual Distress Scale-Revised (FSDS-R) questionnaire consists of 13 items scored on a five-point scale (0, never; 1, rarely; 2, occasionally; 2, frequently; 4, always). The total score is obtained by summing all of the items. Total score ranges from 0 to 52. A higher score corresponds to a greater sexual dysfunction.
Amelioration of the vaginal maturation (VM) index | From baseline to 12 weeks of treatment
  Amelioration of VMI in postmenopausal women in Hyalo Gyn gel group compared to no-treatment group. Vaginal maturation (VM) index is calculated quantifying the percentages of parabasal, intermediate, and superficial cells. The following formula is used: VMI = [1(% superficial cells)] + [0.6(% intermediate cells)] + [0.2(% parabasal cells)]. The index ranges from 0% to 100%.The higher the maturation index, the higher the number of mature cells (0%-49%, low stimulation of the vaginal epithelium; 50%-64%, moderate stimulation of the vaginal epithelium; 65%-100%, high stimulation of the vaginal epithelium).
Patient's global assessment of overall satisfaction | 4 and 12 weeks of treatment
  Patient's global assessment of overall satisfaction in postmenopausal women in Hyalo Gyn gel group compared to no-treatment group.Patient's global assessment (PTGA) is evaluated as the patient's overall satisfaction of the treatment scored on a four grade scale, ranging from 0 to 3 (0= dissatisfied or very dissatisfied, 1= moderately satisfied or satisfied, 2= very satisfied and 3= greatly satisfied). A higher score corresponds to a greater satisfaction.
Ease in the method of Hyalo Gyn gel administration | 4 and 12 weeks of treatment
  Ease in the method of Hyalo Gyn gel administration will be reported by the patients as excellent, good, acceptable, bad or unacceptable
Local tolerability at the application site | 4 and 12 weeks of treatment
  Local tolerability of Hyalo Gyn gel at the application site will be evaluated by both the clinician and the patient through a 5-point scale: 5 = excellent (no reaction), 4 = good (small reaction that spontaneously resolves), 3 = moderate (reaction tolerated with difficulty by the subject), 2 = poor (reaction needing interruption of treatment), 1 = bad (serious reaction)
Safety of the treatment: Collection of adverse events | 4 and 12 weeks of treatment
  Collection of adverse events emerged as consequence of the product application and any other adverse event occurred during the study

CONTACTS AND LOCATIONS:
Locations (2):
- Slovakia (2):
  - Gynkomed s.r.o., Bratislava
  - ULMUS, s r.o., Hlohovec